CLINICAL TRIAL: NCT03716713
Title: CeraShield™ Endotracheal Tube Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: N8 Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N8-2018-02
Record Dates: First submitted 2018-10-19; First posted 2018-10-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CeraShield Endotracheal Tube (Experimental): Subjects who are expected to require mechanical ventilation for 24 hours or longer will be intubated with the CeraShield ETT.
  Interventions: Device: CeraShield Endotracheal Tube

INTERVENTIONS:
Device: CeraShield Endotracheal Tube — Subjects requiring mechanical ventilation with be intubated with the CeraShield ETT

SUMMARY:
Single-arm, feasibility study to evaluate the Ceragenin Coated Endotracheal Tube (the CeraShield ETT) in adults who require intubation and are expected to be mechanically ventilated for ≥ 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older;
* Patients requiring a 7.0mm, 7.5mm, 8.0mm or 8.5mm endotracheal tube;
* Expected to be mechanically ventilated for ≥24 hours.

Exclusion Criteria:

* Currently participating in another clinical trial which conflicts with this trial's design.
* Patients with a pre-existing respiratory infection, i.e., pneumonia.
* Patients with pulmonary contusions.
* Patients with cystic fibrosis.
* Patients demonstrating symptoms of bronchiectasis.
* Patients demonstrating symptoms of severe or massive hemoptysis. Severe or massive hemoptysis defined as greater than 500 ml of blood per day, or greater than 200 ml in six hours.
* Patients who have been intubated within the last 30 days requiring reintubation.
* Women of child-bearing potential who have not undergone a pregnancy test will be excluded from the study.
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 30 days post enrollment or hospital discharge, whichever comes first
  The safety of the CeraShield ETT tube will be assessed by reviewing adverse events in all patients enrolled in the study

SECONDARY OUTCOMES:
Positive QEA | 10 days post intubation
  Determine the incidence of subjects with positive QEA in the patients intubated ≥ 24 hours
Positive ETT colonization | 10 days post intubation
  Determine the incidence of subjects with ETT colonization in the patients intubated ≥ 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided